CLINICAL TRIAL: NCT04815512
Title: Hepatorenal Dysfunctions Among Workers Exposed To Petroleum Products
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abdelsamee Mohammed Ali, lecturer of Occuational and Environmental Medicine, Assiut University
Other Study IDs: HRDs in petroleum workers
Record Dates: First submitted 2021-03-15; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Petroleum Product Toxicity
MeSH Terms: interventions — Liver Function Tests; Kidney Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed group: workers in The Petroleum Pipelines Company who are occupationally exposed to petroleum products will be included in the study.
  Interventions: Diagnostic Test: Liver function tests.; Diagnostic Test: kidney function tests
- Comparison group (control group): healthy administrative workers in assiut university
  Interventions: Diagnostic Test: Liver function tests.; Diagnostic Test: kidney function tests

INTERVENTIONS:
Diagnostic Test: Liver function tests. — serum alanine amino transferase (ALT), aspartate amino transferase (AST), albumin (ALB), alkaline Phosphatase (ALP), total bilirubin.
Diagnostic Test: kidney function tests — creatinine , urea and serum uric acid will be analysed in the serum.

SUMMARY:
The aim of this study is to assess the liver and renal functions of individuals who are occupationally exposed to petroleum products.

DETAILED DESCRIPTION:
Certain peoples have a greater risk of exposure to gasoline vapors; these include filling-station workers, service station attendants, drivers of gasoline trucks and refinery workers.Benzene is metabolized in the liver by cytochrome P450 (CYP) 2E1 to benzene oxide. The metabolites undergo further metabolism through oxidation, dehydrogenation or conjugation with sulfate or glucuronic acid . Activation of benzene and its reactive metabolites leads to continuous production of reactive oxygen species (ROS), which leads to lipid peroxidation and damages DNA, RNA, leading to genetic modification and alterations in the functions of important enzymes (i.e. liver) and proteins .

Volatile organic compounds such as gasoline and other fuels are associated with a wide variety of deleterious health effects including liver and kidney diseases. A comparative cross sectional study was conducted from January 2018 to April 2018 at Mekelle city, Tigray region, Northern Ethiopia among gasoline station workers and reporting that the mean level of ALT, AST, Urea, creatinine, and uric acid was significantly higher among gasoline stations workers when compared to control study participants and there was also a significant increase in ALT, AST, Urea, creatinine and uric acid among gasoline stations with increase duration of exposure .

ELIGIBILITY:
Inclusion Criteria:

for exposed group:

* Apparently health workers who exposed for petroleum products in The Petroleum Pipelines Company in assiut will be included in the study

Exclusion Criteria:

for exposed and Comparison groups

* history of hepatic and renal health problem
* history of taking medications affecting liver and renal function tests

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: workers who are occupationally exposed to petroleum products in The Petroleum Pipelines Company in assiut.The Petroleum Pipelines Company is responsible for transporting and storing crude oil and its products and has a large network of lines.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
measurement of serum alanine amino transferase (ALT) in study participants. | 6 months
  Number of participants with abnormal findings in serum alanine amino transferase (ALT) will be reported.
measurement of serum aspartate amino transferase (AST) in study participants. | 6 months
  Number of participants with abnormal findings in serum aspartate amino transferase (AST) will be reported.
measurement of serum total bilirubin in study participants. | 6 months
  Number of participants with abnormal findings in serum total bilirubin will be reported.
measurement of serum albumin (ALB) in study participants. | 6 months
  Number of participants with abnormal findings in serum albumin (ALB) will be reported.

SECONDARY OUTCOMES:
Measurement of serum urea in study participants. | 6 months
  Number of participants with abnormal findings in serum urea will be reported.
Measurement of serum Creatinine in study participants. | 6 months
  Number of participants with abnormal findings in serum Creatinine will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan M. Ahmed, Prof., Study Chair — Assiut University

REFERENCES:
- [Background] Malini SS, Maithily K. Analysis of oxidative stress in chronic exposure to petroleum hydrocarbons in Karnataka,India. Asia Pac J Med Toxicol. 2017; 6(1):6-11.
- [Background] Bin-Mefrij M, Alwakeel S. The effect of fuel inhalation on the kidney and liver function and blood indices in gasoline station workers. Adv Nat Appl Sci. 2017; 11(1):45-50.
- [Background] Olmedo-Buenrostro BA, Ortega-Ortiz JG, Guzman-Esquivel J, Delgado-Enciso OG, Ceja-Espiritu G,Paz-Michel BA, et al. Workplace gasoline exposure increases the risk for early renal dysfunction: A case-control study in Mexico. Biomed Res. 2017; 28 (22): 9859-9863.
- [Background] Asefaw T, Wolde M, Edao A, Tsegaye A, Teklu G, Tesfay F, Gebremariam G. Assessment of liver and renal function tests among gasoline exposed gas station workers in Mekelle city, Tigray region, Northern Ethiopia. PLoS One. 2020 Oct 9;15(10):e0239716. doi: 10.1371/journal.pone.0239716. eCollection 2020. PMID 33035217